CLINICAL TRIAL: NCT00159315
Title: Adenosine 5'-Triphosphate (ATP) Challenge in Healthy Non-smokers, Current Smokers and Patients With Mild Asthma and Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: ATP/AMP Challenge in Healthy Non-smokers, Smokers, Patients With Asthma, and Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Duska Scientific Co. (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DHTABPT0336
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Asthma; COPD; Smoking
Keywords: Healthy Volunteers (smokers); Healthy Volunteers (Non-smokers); Asthma Patients; COPD Patients
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Smoking | interventions — Adenosine Triphosphate; Adenosine Monophosphate

ARMS (2):
- Nebulised ATP (Experimental)
  Interventions: Procedure: Inhalation Challenge with ATP; Procedure: Inhalation Challenge with AMP
- Inhaled Adenosine (Active Comparator)
  Interventions: Procedure: Inhalation Challenge with ATP; Procedure: Inhalation Challenge with AMP

INTERVENTIONS:
Procedure: Inhalation Challenge with ATP
Procedure: Inhalation Challenge with AMP

SUMMARY:
In this randomised, cross-over, controlled study, a total of 84 subjects will be included: 12 healthy non-smoking volunteers; 12 current smokers; 30 patients with mild steroid-naïve asthma; and 30 patients with mild-moderate COPD.

Each subject will have 1 screening visit (if necessary) and 2 study visits. At visits 2 and 3 the effects of adenosine 5'-triphosphate (ATP) or adenosine 5'-monophosphate (AMP) challenge, given in a random order, will be tested.

DETAILED DESCRIPTION:
Background: Extracellular adenosine 5'-triphosphate (ATP) stimulates vagal C and Aδ fibers in the lung, resulting in pronounced bronchoconstriction and cough mediated by P2X2/3 receptors located on vagal sensory nerve terminals. We investigated the effects of nebulized ATP on cough and symptoms in control subjects, healthy smokers, and patients with COPD and compared these responses to the effects of inhaled adenosine, the metabolite of ATP.

Methods: We studied the effects of inhaled ATP and adenosine monophosphate (AMP) on airway caliber, perception of dyspnea assessed by the Borg score, cough sensitivity, and ATP in exhaled breath condensate in healthy nonsmokers (n = 10), healthy smokers (n = 14), and patients with COPD (n = 7).

Results: In comparison with healthy subjects, ATP induced more dyspnea, cough, and throat irritation in smokers and patients with COPD, and the effects of ATP were more pronounced than those of AMP. The concentration of ATP in the exhaled breath condensate of patients with COPD was elevated compared with that of healthy subjects.

Conclusions: Smokers and patients with COPD manifest hypersensitivity to extracellular ATP, which may play a mechanistic role in COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy non-smokers (n=12)

   * Normal spirometry
   * Forced expiratory volume in 1 second (FEV1) reversibility of < 15% after inhaled beta2-agonists*
2. At risk (current smokers) (n=12)*

   * Normal spirometry, chronic symptoms (cough, sputum production)
   * FEV1 reversibility of < 15% after inhaled beta2-agonists* (* = Global Strategy for the Diagnosis, Management, and Prevention of COPD)
3. Mild steroid-naïve asthma (n=30)

   * FEV1 more than or equal to 80%
4. Mild-moderate COPD (n=30)

   * FEV1 50-80%

Exclusion Criteria:

1. Pregnancy, breast-feeding, or planned pregnancy during the study.
2. Fertile women not using acceptable contraceptive measures, as judged by the investigator
3. Upper respiratory infection within the last 4 weeks
4. Subjects who have received research medication within the previous one month
5. Subjects unable to give informed consent
6. Any psychiatric condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-10 (Actual); Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
PC20 of ATP and AMP | On administration
  PC20 of ATP and AMP
Lung function | On administration
  Spirometry
Borg score | On administration
  Measurement of DYSPNEA
Impulse oscillometry (IOS) | On administration
  Small airway function

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Result] Basoglu OK, Barnes PJ, Kharitonov SA, Pelleg A. Effects of Aerosolized Adenosine 5'-Triphosphate in Smokers and Patients With COPD. Chest. 2015 Aug;148(2):430-435. doi: 10.1378/chest.14-2285. PMID 25590209